CLINICAL TRIAL: NCT00204178
Title: The Role of Reactive Oxygen Species in Ischaemia-Reperfusion Injury of the Transplanted Kidney
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Uniwersytet Mikolaja Kopernika w Toruniu (Other)
Other Study IDs: KB/38/2003
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-12-01 (Estimated); Status verified 2005-08

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplantation; Reperfusion injury
MeSH Terms: conditions — Reperfusion Injury | interventions — Oxidative Stress

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Behavioral: Oxidative stress in kidney transplant recipients

SUMMARY:
Measurement of reactive oxygen species production and antioxidant system status before and directly after reperfusion of the transplanted kidney and influence of oxidant stress on kidney function in 2 and 6 weeks.

DETAILED DESCRIPTION:
Oxidative stress is one of the most important factors in ischaemia-reperfusion injury to the transplanted organ. In kidney transplant recipients following factors were measured: glutathione level, activities of glutathione peroxidase (GSH-PX), catalase (CAT) and superoxide dismutase (SOD) and superoxide anion production by granulocytes in whole blood without and after the stimulation with zymosan.

Blood was sampled from peripheral vein (before reperfusion) and directly from renal vein (5 and 15 minutes after reperfusion).

Transplanted kidney function was evaluated by the incidence and length of Delayed Graft Function and serum creatinine level in 2 and 6 weeks after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients accepted for and undergoing cadaveric kidney transplantation

Exclusion Criteria:

* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-04; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Zbigniew Wlodarczyk, MD,PhD, Study Director — Klinika Transplantologii Collegium Medicum UMK w Toruniu
Locations (1):
- Klinika Transplantologii, Szpital Uniwersytecki, ul. M. Sklodowskiej-Curie 9, Bydgoszcz, Poland